CLINICAL TRIAL: NCT01390545
Title: VELVET (Veltuzumab Various Doses Exploratory Trial), a Randomized, Double Blind, Placebo Controlled, Multicentre, Multinational Phase II Dose Range Finding Trial in Subjects With Moderate to Severe Rheumatoid Arthritis Insufficiently Controlled With Either Methotrexate Alone or Methotrexate Plus Anti-tumour Necrosis Factor Biological Treatment, Comparing 3 Different Subcutaneous Dosages of Anti-CD20 Monoclonal Antibody Veltuzumab to Placebo as an add-on Therapy to Methotrexate.
Brief Title: VELVET, a Dose Range Finding Trial of Veltuzumab in Subjects With Moderate to Severe Rheumatoid Arthritis
Acronym: VELVET
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial re-design; no safety issues identified
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VT-4001-001-SP; 2010-022378-15 (EudraCT Number); U1111-1136-3415 (Registry Identifier: WHO)
Record Dates: First submitted 2011-07-05; First posted 2011-07-11 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; anti-CD20 antibody; subcutaneous
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — veltuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Veltuzumab 80 mg (Active Comparator)
  Interventions: Drug: Veltuzumab
- Veltuzumab 160 mg (Active Comparator)
  Interventions: Drug: Veltuzumab
- Veltuzumab 320 mg (Active Comparator)
  Interventions: Drug: Veltuzumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Veltuzumab

INTERVENTIONS:
Drug: Veltuzumab — administered once weekly (days 1, 8, 15 and 22) by subcutaneous injection

SUMMARY:
This is a multi-national, multi-centre, placebo-controlled, double-blind, randomized, 4-arm parallel group trial, comparing three different dose levels (80 mg, 160 mg and 320 mg) of veltuzumab to placebo, administered weekly (days 1, 8, 15 and 22) by subcutaneous (sc) injection to subjects with moderate to severe rheumatoid arthritis (RA) (cumulative veltuzumab doses 320 mg, 640 mg, and 1280 mg, respectively). All subjects will be on continued stable co-medication with methotrexate (MTX).

DETAILED DESCRIPTION:
The trial comprises a screening phase (4 to 12 weeks prior to first administration of veltuzumab), a 4-week treatment phase (weeks 1 to 4), a core phase from week 4 to week 24, and a follow-up phase from week 24 to week 48. The primary end-point, the American College of Rheumatology 20 (ACR 20) response rate, will be evaluated at week 24.

The objectives of this trial are:

* To investigate the efficacy, safety and tolerability at week 24 of three different sc dose levels of the humanized anti-CD20 antibody veltuzumab as an add-on treatment to MTX compared to MTX alone in subjects with moderate to severe RA
* To evaluate the durability of the clinical response and safety of veltuzumab over 48 weeks
* To identify the dosage(s) of veltuzumab with the most favourable benefit-risk profile to be further evaluated in the subsequent phase II/III clinical program in subjects with moderate to severe RA.

Current status of the trial: Following the voluntary temporary halt of the VELVET dose range finding trial, the sponsor has decided to redesign the protocol and start a new trial as soon as possible.

All patients treated prior to the voluntary halt have completed their safety assessments. It was decided to terminate the VELVET trial and consequently not to recommence enrollment.

In the VELVET trial, a total of 11 patients received trial medication prior to the voluntary temporary halt. No efficacy conclusions according to protocol can be drawn from the 11 patients treated. Based on the collected clinical data from this trial, there is no clinical safety signal and no increased clinical safety risk observed to date that precludes continued clinical investigation of veltuzumab.

ELIGIBILITY:
Main Inclusion Criteria:

* Active disease defined as:

  * Diagnosis of RA using the ACR criteria for the classification of RA for at least 6 months prior to trial entry (Screening, Visit 1)
  * Swollen joint count (SJC) ≥ 6 and tender joint count (TJC) ≥ 6 referred to as the 66/68 - joint count system
  * High sensitivity C-reactive protein (hs-CRP) ≥ 15 mg/L and/or an erythrocyte sedimentation rate (ESR) ≥ 28 mm/hour
  * Positive rheumatoid factor (RF) ≥ 14 IU/mL and/or anti-cyclic citrullinated protein (CCP) ≥ 20 U
* An inadequate response (insufficient initial or loss of response and/or intolerance to at least one administration of these agents) to previous or current treatment with either MTX alone or MTX plus anti-tumour necrosis factor alpha (anti-TNFα) biological treatment. Subjects should not have received more than two different anti-TNFα therapies.
* Receiving MTX 15-25 mg/week (oral or parenteral) for at least 20 weeks, including the last 6 weeks prior to Baseline (Visit 3, Day 1) at a stable dose via the same route of administration and formulation. A stable dose of 12.5 mg of MTX is acceptable if the MTX dose has been reduced for reasons of toxicity, e.g. pulmonary, hepatic or haematological toxicity. MTX co-medication will be continued until the end of the trial (Week 48)

Main Exclusion Criteria:

* Primary or secondary immunodeficiency including HIV infection
* Evidence of acute or chronic infection with hepatitis B and C virus (HBV and HCV)
* Evidence (e.g. chest X-ray [posterior-anterior view], tuberculin/ PPD skin test, etc., according local guidelines) and/or history of active tuberculosis (TB), prior to successfully completing an anti-TB treatment. X-rays performed prior to inclusion (Screening, Visit 1) into the trial are accepted provided they were done within 3 months prior to Screening (Visit 1). Subjects with latent TB infection (LTBI) can be included
* Significant cardiac disease or history of severe COPD
* Diabetes mellitus type 1 or unstable type 2
* History of cancer within the last 5 years treated with anti-cancer chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
American College of Rheumatology 20 (ACR20) response rate at completion of week 24 | 24 weeks
  ACR20 response rate is defined as improvement from baseline to endpoint fulfilling the following criteria:
  * ≥ 20 percent reduction in the Tender joint count (TJC) (66/68 joint count system)
  * ≥ 20 percent reduction in the Swollen joint count (SJC) (66/68 joint count system)
  * ≥ 20 percent reduction in three of the following additional measures:
    * Patient's assessment of pain
    * Patient's global assessment of disease activity
    * Physician's global assessment of disease activity
    * Degree of disability
    * Level of acute-phase reactant (CRP)

SECONDARY OUTCOMES:
ACR50/70 response rate | 24 and 48 weeks
  ACR50/70 response rate is defined as improvement from baseline to endpoint fulfilling the following criteria:
  * 50/70 percent reduction in the TJC (66/68 joint count system)
  * 50/70 percent reduction in the SJC (66/68 joint count system)
  * 50/70 percent in three of the following additional measures:
    * Patient's assessment of pain
    * Patient's global assessment of disease activity
    * Physician's global assessment of disease activity
    * Degree of disability
    * Level of acute-phase reactant (CRP)
ACR20 response rate | 48 weeks
  ACR20 response rate is defined as improvement from baseline to endpoint fulfilling the following criteria:
  * 20 percent reduction in the TJC (66/68 joint count system)
  * 20 percent reduction in the SJC (66/68 joint count system)
  * 20 percent reduction in three of the following additional measures:
    * Patient's assessment of pain
    * Patient's global assessment of disease activity
    * Physician's global assessment of disease activity
    * Degree of disability
    * Level of acute-phase reactant (CRP)
Further efficacy analyses (Hybrid ACR response, DAS28-CRP, EULAR response) | 24 and 48 weeks
  To further demonstrate efficacy of veltuzumab

CONTACTS AND LOCATIONS:
Locations (57):
- United States (8):
  - Nycomed Investigational Site, La Mesa, California
  - Nycomed Investigational Site, Los Angeles, California
  - Nycomed Investigational Site, Upland, California
  - Nycomed Investigational Site, Aventura, Florida
  - Nycomed Investigational Site, Las Vegas, Nevada
  - Nycomed Investigational Site, Charleston, South Carolina
  - Nycomed Investigational Site, Nashville, Tennessee
  - Nycomed Investigational Site, San Antonio, Texas
- Argentina (5):
  - Nycomed Investigational Site, Caba, Buenos Aires
  - Nycomed Investigational Site, Córdoba, Córdoba Province
  - Nycomed Investigational Site, San Juan, San Juan Province
  - Nycomed Investigational Site, Santa Fe, Santa Fe Province
  - Nycomed Investigational Site, San Miguel de Tucumán, Tucumán Province
- Canada (7):
  - Nycomed Investigational Site, Calgary, Alberta
  - Nycomed Investigational Site, Kitchener, Ontario
  - Nycomed Investigational Site, Ottawa, Ontario
  - Nycomed Investigational Site, St. Catharines, Ontario
  - Nycomed Investigational Site, Toronto, Ontario
  - Nycomed Investigational Site, Windsor, Ontario
  - Nycomed Investigational Site, Saskatoon, Saskatchewan
- Czechia (6):
  - Nycomed Investigational Site, Hlučín
  - Nycomed Investigational Site, Hostivice
  - Nycomed Investigational Site, Pilsen
  - Nycomed Investigational Site, Prague
  - Nycomed Investigational Site, Uherské Hradiště
  - Nycomed Investigational Site, Zlín
- Germany (2):
  - Nycomed Investigational Site, Bad Nauheim
  - Nycomed Investigational Site, Würzburg
- Hungary (7):
  - Nycomed Investigational Site, Debrecen
  - Nycomed Investigational Site, Kecskemét
  - Nycomed Investigational Site, Kiskunhaias
  - Nycomed Investigational Site, Kistarcsa
  - Nycomed Investigational Site, Mezőkövesd
  - Nycomed Investigational Site, Székesfehérvár
  - Nycomed Investigational Site, Szolnok
- Italy (4):
  - Nycomed Investigational Site, Arenzano (GE)
  - Nycomed Investigational Site, Jesi (AN)
  - Nycomed Investigational Site, Massa
  - Nycomed Investigational Site, Valeggio S/M (VR)
- Mexico (7):
  - Nycomed Investigational Site, Guadalajara, Jalisco
  - Nycomed Investigational Site, Distrito Federal, Mexico
  - Nycomed Investigational Site, Distrito Federal, México
  - Nycomed Investigational Site, Monterrey, Nuevo León
  - Nycomed Investigational Site, Culiacán, Sinaloa
  - Nycomed Investigational Site, Mazatlán, Sinaloa
  - Nycomed Investigational Site, Ciudad Obregón, Sonora
- Poland (6):
  - Nycomed Investigational Site, Bialystok
  - Nycomed Investigational Site, Bydgoszcz
  - Nycomed Investigational Site, Lublin
  - Nycomed Investigational Site, Poznan
  - Nycomed Investigational Site, Sopot
  - Nycomed Investigational Site, Warsaw
- Spain (3):
  - Nycomed Investigational Site, Seville, Andalusia
  - Nycomed Investigational Site, Barakaldo, Basque Country
  - Nycomed Investigational Site, A Coruña, Galicia
- United Kingdom (2):
  - Nycomed Investigational Site, Ashford, Middlesex
  - Nycomed Investigational Site, Barnsley, S. Yorkshire